CLINICAL TRIAL: NCT00382889
Title: Multinational, Double Blind, Randomised, Parallel Group Study on the Therapeutic Efficacy and Safety of Beclomethasone Dipropionate 250 mg Combined With Salbutamol 100 mg in the Treatment of Patients With Mild Persistent Asthma.
Brief Title: As Needed Beclomethasone/Salbutamol Combination in Single Inhaler for Mild Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MC/PR/1401/001/01
Record Dates: First submitted 2006-09-29; First posted 2006-10-02 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Asthma
Keywords: Anti-Asthmatic Agents; corticosteroids; symptom-driven; beclomethasone; salbutamol
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; Albuterol

INTERVENTIONS:
Drug: beclomethasone/salbutamol combination
Drug: beclomethasone
Drug: salbutamol

SUMMARY:
The aim of this study is to reveal that inhaled corticosteroid therapy combined with a short-acting beta2- agonist given on a symptom driven basis is as effective as traditional asthma therapy.

Thus, three advantages will be achieved:

1. better compliance with treatment since patients will most likely have to administer the treatment less frequently,
2. maximum pharmacological effect with the least amount of drug and
3. less economic burden on health care providers.

DETAILED DESCRIPTION:
Asthma is widely recognised as a chronic inflammatory disorder of the airways. The 1997 American National Heart Lung and Blood Institute (NHLBI) Guidelines states that a firm scientific basis exists to indicate that asthma results from complex interactions among inflammatory cells, mediators and the cells and tissues resident in the airways.

Despite the existence of effective therapy people still die from asthma. It is pertinent to state that the clinical effect of a drug is not only dependent on the specific action of the drug, but also on the patient's way of using it. Therefore, compliance is an important factor especially for chronic disorders such as asthma. Indeed, non compliance with asthma therapy is a serious problem. It has been reported that drug side effects, lifestyle, social and economic factors, method of drug delivery and dosing are factors that contribute to poor compliance. The consequences of poor compliance lead to increased morbidity due to increased symptoms and asthma exacerbation.

The NHLBI Guidelines recommend daily treatment for patients with mild persistent asthma with inhaled glucocorticoids (200-500mcg/die) and short-acting bronchodilators as needed but no more than 3-4 times a day.

Comparisons: beclomethasone dipropionate 250 mg combined with salbutamol 100 mg "as needed", vs salbutamol 100 mg alone "as needed", vs beclomethasone 250 mg twice a day plus salbutamol 100 mg "as needed" and vs beclomethasone dipropionate 250 mg combined with salbutamol 100 mg twice a day plus salbutamol 100 mg "as needed", in the treatment of patients with mild persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild persistent asthma as defined by NHLBI/WHO 97; for at least 6 months;
* FEV1 ³ 75% of predicted normal value;
* Positive response to the reversibility test to b2 agonist, defined as an increase > 12% in the FEV1 measured 30 minutes following 2 puffs (2x100mg) of inhaled Salbutamol spray, or positive methacholine challenge (PC20<8mg/ml or PD20<1 mg) within the previous 6 months;
* Stable asthma. Asthma is defined stable if none of the following occurred during the last 14 days of the run-in period: diurnal variation of more than 20% in PEF on 2 consecutive days; use of four or more inhalations of b2 agonist per day on two consecutive days; need the use of oral corticosteroids;

Exclusion Criteria:

* COPD as defined by the ERS - Consensus Statement;
* Patients with more than 10 packs/year of cigarettes history and current smokers;
* History of near fatal asthma and/or admission in intensive care unit because of asthma;
* One severe exacerbation during the run-in period;
* Three or more courses of oral corticosteroids or hospitalisation for asthma during the previous 1 year;
* Patients treated with more than 500 mcg/day of beclomethasone or equivalent for more than 6 months in the previous last year;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480
Dates: Start 2002-08; Study Completion 2004-09

PRIMARY OUTCOMES:
The primary outcome for comparison across treatment groups was the mean value of morning PEF measured during the last 2 weeks of treatment (weeks 23-24)

SECONDARY OUTCOMES:
Number of exacerbations
Time to first severe exacerbation
Improvement of asthma symptoms (symptom scores)
Need for short acting b2 agonists
Variation of respiratory parameters (FEV1, PEF, FVC, FEV1/FVC, FEF25-75) immediately before and 30 min after a test with a short-acting b2 agonist
evening PEF
Diurnal variability of PEF
Nocturnal asthma (nocturnal awakening because of asthma)
Nights and days without asthma symptoms (score 0)

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo M Fabbri, MD, Principal Investigator — Clinica di Malattie dell'Apparato Respiratorio, Dipartimento di Oncologia, Ematologia e Pneumologia, Università di Modena e Reggio Emilia, Italy
Locations (25):
- Austria (2):
  - Ambulance for pediatrics and Pneumology, Vienna
  - Pulmologisches Zentrum Der Stadt Wien, Vienna
- Italy (9):
  - Dip. di Pneumologia - Osp. Tommaselli, Catania
  - Nuove Cliniche Arcispedale S.Anna, Ferrara
  - DIMI - Dip. Medicina Interna - Univ. di Genova - clinica di malattie apparato respiratorio e allergologico, Genova
  - Dipartimento di scienze mediche oncologiche e radiologiche - sez. malattie apparato respiratorio, Modena
  - Univ. di Padova - Dipartimento di medicina ambientale e sanità pubblica, Padua
  - Istituto di Fisiopatologia Respiratoria CNR - Ospedale Cervello, Palermo
  - Clinica Pneumologica padiglione Rasori - Univ. di Parma, Parma
  - Clinica di Malattie dell'Apparato Respiratorio dell'Univ. di Pavia - Policlinico S. Matteo, Pavia
  - Reparto Fisiologia Respiratoria - dip. Cardiotoracico - Ospedale Cisanello, Pisa
- Poland (11):
  - Outpatient Clinic of Internal Diseases and Allergology, Bialystok
  - Specialist Group Medex, Bielsko-Biala
  - Clinic of Internal Diseases Atopia Al., Krakow
  - Pulmonologic Clinic - Poludnie os. Krakowiakòw, Krakow
  - Clinic of Pneumology and Allergology, Lòdz
  - Clinic of Tubercolosis and Lung Diseases, Lòdz
  - Clinic of Pneumology - Institute of Internal Medicine of Medical Academy, Lódz
  - Institute of Occupational Medicine - Clinic of Occupational Disesase, Lódz
  - Clinic of Infection Diseases and Allergology - Central Clinical Hospital of Military Medical Academy, Warsaw
  - Clinic of Pneumology and Allergology A.M., Warsaw
  - Clinic of Pneumology and Allergology of Medical Academy, Warsaw
- Spain (3):
  - Hospital Vall d'Hebron de Barcelona, Barcelona
  - H.General de Vic, Servicio de Neumologia, Barcelona
  - Hospital de Matarò, Mataró

REFERENCES:
- [Result] Papi A, Canonica GW, Maestrelli P, Paggiaro P, Olivieri D, Pozzi E, Crimi N, Vignola AM, Morelli P, Nicolini G, Fabbri LM; BEST Study Group. Rescue use of beclomethasone and albuterol in a single inhaler for mild asthma. N Engl J Med. 2007 May 17;356(20):2040-52. doi: 10.1056/NEJMoa063861. PMID 17507703